CLINICAL TRIAL: NCT04647721
Title: Evaluation of the Effectiveness and Safety of Radiesse for the Correction of Moderate to Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Merz North America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: M900311009
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Results first posted 2023-01-23 (Actual); Last update posted 2023-01-23 (Actual); Status verified 2023-01

CONDITIONS: Correction of Moderate to Severe Nasolabial Folds (NLFs)

STUDY DESIGN:
Intervention Model Description: Split-face
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Left side Radiesse® / Right side Restylane® (Experimental)
  Interventions: Device: Radiesse injectable implant (dermal filler); Device: Restylane injectable implant (dermal filler)
- Left side Restylane® / Right side Radiesse® (Experimental)
  Interventions: Device: Radiesse injectable implant (dermal filler); Device: Restylane injectable implant (dermal filler)

INTERVENTIONS:
Device: Radiesse injectable implant (dermal filler) — Subdermal injection.
  Other Names: Calcium hydroxylapatite particles suspended in an aqueous based gel carrier.
Device: Restylane injectable implant (dermal filler) — Subdermal injection.
  Other Names: Hyaluronic acid

SUMMARY:
Effectiveness: The purpose of this study is to demonstrate the non-inferiority of Radiesse (CaHA) to Restylane (HA) following subdermal implantation for the correction of moderate to severe facial wrinkles and folds, such as NLFs.

Safety: To evaluate the incidence and type of adverse events and serious adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Has symmetrical NLFs, with the same WSRS score of 3 or 4 (moderate or severe) for both right and left NLFs, as determined on live assessment by the blinded evaluator.
* Is ≥ 22 and ≤ 65 years of age.
* Is willing to abstain from all other aesthetic treatments on any part of the face, including but not limited to injectable fillers, implants, neurotoxin, skin peels, laser treatments, surgical treatments, etc. for the trial's duration.

Exclusion Criteria:

* Has an acute inflammatory process or active infection at the injection site.
* Has received mid- and/or lower-facial region treatments with any dermal fillers.
* Has received facial dermal therapies.
* Had prior surgery in the mid- and/or lower-facial area, including the NLFs, or has a permanent implant or graft in the mid- and/or lowerfacial area that could interfere with effectiveness assessments.

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2022-04-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Merz Medical Expert, Study Director — Merz North America, Inc.
Locations (7):
- China (7):
  - Peking University First Hospital, Merz Investigational Site #0860003, Beijing
  - Peking University Third Hospital, Merz Investigational Site #0860009, Beijing
  - The Third Affiliated Hospital, Sun Yat-Sen University, Merz Investigational Site #0860023, Guangzhou
  - Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Merz Investigational Site #0860030, Hangzhou
  - Zhejiang Provincial People's Hospital, Merz Investigational Site #0860005, Hangzhou
  - Zhongda Hospital Southeast University, Merz Investigational Site #0860022, Nanjing
  - RenMin Hospital of Wuhan University, Merz Investigational Site #0860014, Wuhan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 7 investigational sites in China.
Pre-assignment Details: Of the 134 enrolled, 13 subjects were exited as screen failures. This reporting group includes all randomized subjects (121).
Units Other Than Participants: Nasolabial Folds (NLFs)
Groups:
- Left Side Radiesse® / Right Side Restylane®; Left Side Restylane® / Right Side Radiesse®: Radiesse injectable implant (dermal filler): Subdermal injection. Restylane injectable implant (dermal filler): Subdermal injection.
Period: Overall Study
Arm/Group | Left Side Radiesse® / Right Side Restylane® | Left Side Restylane® / Right Side Radiesse®
Started | 61; 122 Nasolabial Folds (NLFs) | 60; 120 Nasolabial Folds (NLFs)
Safety Population (1 subject randomized to Left side Restylane® / RIght side Radiesse® did not receive any treatment and was excluded from the safety population.) | 61; 122 Nasolabial Folds (NLFs) | 59; 118 Nasolabial Folds (NLFs)
Completed | 59; 118 Nasolabial Folds (NLFs) | 58; 116 Nasolabial Folds (NLFs)
Not Completed | 2; 4 Nasolabial Folds (NLFs) | 2; 4 Nasolabial Folds (NLFs)
Not completed — Withdrawal by Subject | 0 | 2
Not completed — Lost to Follow-up | 2 | 0

BASELINE CHARACTERISTICS:
Population: This analysis population includes all randomized subjects who received investigational product at least once (Safety Population).
Groups:
- Radiesse and Restylane: Subjects were randomized to receive Radiesse in either of the two nasolabial folds and Restylane in the respective other.
Arm/Group | Radiesse and Restylane
Number analyzed (Participants) | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.6 (9.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 120
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 24 on the Wrinkle Severity Rating Scale (WSRS)
Description: Severity of the nasolabial folds (NLFs) was assessed and measured using the 5-point Wrinkle Severity Rating Scale (WSRS), where 1=absent and 5=extreme. A lower score indicates better outcome.
Time Frame: Baseline and Week 24 after last injection, up to 28 weeks
Population: This analysis population includes all randomized and treated subjects with no major protocol deviations or other events that impact analysis of the primary effectiveness endpoint (Per Protocol Set) with observed cases at the Week 24 visit.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: NLFs
Groups:
- Restylane: Restylane injectable implant (dermal filler): Subdermal injection.
- Radiesse: Radiesse injectable implant (dermal filler): Subdermal injection.
Arm/Group | Restylane | Radiesse
Number analyzed (Participants) | 115 | 115
Number analyzed (NLFs) | 115 | 115
score on a scale
  Baseline | 3.4 (0.50) | 3.4 (0.50)
  Week 24: number analyzed (Participants) | 114 | 114
  Week 24: number analyzed (NLFs) | 114 | 114
  Week 24 | 2.4 (0.62) | 2.4 (0.70)
Statistical Analysis 1: Comparison: Restylane vs Radiesse; Test type: Non-Inferiority — Non-inferiority margin of 0.5. The two-sided 95% confidence interval (CI) for the treatment difference was constructed using the repeated-measures analysis of covariance (ANCOVA); Difference in Least Squares Means = 0.03, 95% CI 2-sided [-0.07 to 0.12]

2. Secondary Outcome: Proportion of Subjects With Improvement on the Investigator Global Aesthetic Improvement Scale (iGAIS) for Each Nasolabial Fold (NLF) at Week 24
Description: The Investigator Global Aesthetic Improvement Scale is a subjective assessment where the treating physician describes the degree of improvement in facial appearance ranging from "Very much improved" (+3) to "Very much worse" (-3). The investigator was asked to rate each NLF separately and select the rating that best applied when asked "What is the overall impression of aesthetic change of the subject's NLF due to treatment, compared to the pretreatment photograph". Improvement was defined as a rating of +1, +2, or +3. The higher the iGAIS score, the greater the improvement. Proportion refers to percentage of participants.
Time Frame: Week 24 after last injection, up to 28 weeks
Population: Subjects in the Per Protocol Set with observed cases at the Week 24 visit.
Measure: Number; unit: percentage of participants
Units Other Than Participants: NLFs
Arm/Group | Restylane | Radiesse
Number analyzed (Participants) | 114 | 114
Number analyzed (NLFs) | 114 | 114
percentage of participants | 77.19 | 77.19
Statistical Analysis 1: Comparison: Restylane vs Radiesse; Test type: Other; Risk Difference (RD) = 0.00, 95% CI 2-sided [-6.35 to 6.35]

3. Secondary Outcome: Proportion of Subjects With Any Improvement on the Subject Global Aesthetic Improvement Scale (sGAIS) for Each Nasolabial Fold (NLF) at Week 24
Description: The Subject Global Aesthetic Improvement Scale is a subjective self-assessment where the subject independently describes the degree of improvement in facial appearance ranging from "Very much improved" (+3) to "Very much worse" (-3). Subjects rated each NLF separately when asked "What is the overall impression of aesthetic change of your NLF due to treatment, compared to the pretreatment photograph?" Improvement is defined as a rating of +1, +2, or +3. The higher the sGAIS score, the greater the improvement. Proportion refers to percentage of participants.
Time Frame: Week 24 after last injection, up to 28 weeks
Population: Subjects in the Per Protocol Set with observed cases at the Week 24 visit.
Measure: Number; unit: percentage of participants
Units Other Than Participants: NLFs
Arm/Group | Restylane | Radiesse
Number analyzed (Participants) | 114 | 114
Number analyzed (NLFs) | 114 | 114
percentage of participants | 80.70 | 82.46
Statistical Analysis 1: Comparison: Restylane vs Radiesse; Test type: Other; Risk Difference (RD) = 1.75, 95% CI 2-sided [-3.08 to 6.74]

4. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (AE) Related to Radiesse
Description: Defined as AEs with onset at or after date of first administration of Radiesse. An AE was considered to be "related" if a causal relationship between Radiesse or the treatment procedure and the AE is at least reasonably possible.
Time Frame: Baseline to week 48 after last injection, up to 52 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Radiesse: Subjects with event related to Radiesse injectable implant(dermal filler)
Arm/Group | Radiesse
Number analyzed (Participants) | 120
Participants | 23

ADVERSE EVENTS:
Time Frame: From first treatment up to the end of study (Week 48 after last injection), an average of 52 weeks
Description: The investigator asked the participant for adverse events (AEs) systematically at each visit. "At Risk" population for Restylane and Radiesse AEs are reported in units of NLFs; Non-NLF population is reported in units of subjects.
Groups:
- Restylane: Events affecting the NLF treated with Restylane
- Radiesse: Events affecting the NLF treated with Radiesse
- Non-NLF: Subjects with events not affecting either of the two NLFs
Arm/Group | Restylane | Radiesse | Non-NLF
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/120 | 0/120
Serious Adverse Events (participants affected / at risk) | 0/120 | 0/120 | 7/120
Other Adverse Events (participants affected / at risk) | 7/120 | 18/120 | 9/120
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Restylane (N=120) | Radiesse (N=120) | Non-NLF (N=120)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 1
Cervical dysplasia (Reproductive system and breast disorders) | 0 | 0 | 1
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Restylane (N=120) | Radiesse (N=120) | Non-NLF (N=120)
Injection site induration (General disorders) | 7 | 15 | 0
Injection site nodule (General disorders) | 4 | 12 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Publication of study information usually requires agreement with the sponsor. In case of justified doubts by the sponsor, the INVESTIGATOR will consider these doubts in the publication as long as the scientific neutrality is not affected.

DOCUMENTS (2):
  • Study Protocol (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT04647721/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT04647721/SAP_001.pdf